CLINICAL TRIAL: NCT01092442
Title: CryoValve SG Pulmonary Human Heart Valve Post Clearance Study
Acronym: SGPV
Status: Completed | Type: Observational
Sponsor: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Organization: CryoLife (Unknown)
Other Study IDs: CSG801.002-M
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Valve Stenosis; Pulmonary Valve Insufficiency; Aortic Valve Stenosis; Aortic Valve Insufficiency
Keywords: Pulmonary Valve; Right Ventricular Outflow Tract Reconstruction; Ross Procedure
MeSH Terms: conditions — Pulmonary Valve Stenosis; Pulmonary Valve Insufficiency; Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective Patients: Retrospective Patients: The patient group who had the CryoValve SG Pulmonary Human Heart Valve implanted prior to the February 2008 clearance of the valve.
  Interventions: Procedure: Echocardiogram
- Prospective Patients: Prospective Patients: The patient group that had the CryoValve SG Pulmonary Human Heart Valve implanted after the February 2008 clearance of the valve.
  Interventions: Procedure: Echocardiogram

INTERVENTIONS:
Procedure: Echocardiogram — Patients will have a yearly echocardiogram after enrollment in the study.

SUMMARY:
The purpose of this study is to collect long-term follow-up data of the CryoValve SG Pulmonary Human Heart Valve.

DETAILED DESCRIPTION:
The CryoValve SG pulmonary human heart valve is recovered from deceased human donors, treated with the SynerGraft® process,which is designed to reduce the donor cells present on the graft. The valve is then cryopreserved for storage until use. Removing cells from the heart valve has been shown to reduce a component of the immune response after implant compared to a standard allograft valve. However, it is not known how this affects the long-term durability of the valve.

ELIGIBILITY:
• Retrospective Patients

o Sequential patients implanted with a CryoValve SG Pulmonary Human Heart Halve as a Ross or RVOT reconstruction between February 2000 and March 2004 who were included in the 510(k) data collection will be identified using the following general criteria to aid in selection of patients who are most likely to provide adequate follow-up data: Patient is alive and the implanted valve is still in place (has not been explanted).

Patient is still under the care of the implanting institution or the implanting surgeon.

Patient was identified as previously providing data for at least one echocardiographic follow-up assessment at a minimum of one year post-implant.

* Additionally, prospective enrolling centers will have the option to enroll retrospective patients. At these centers, all consecutive patients identified from valve implant data at CryoLife, implanted with a CryoValve SG Pulmonary Valve as a valved pulmonary valve prior to Clearance in 2008 will be targeted for inclusion in the retrospective patient data collection.

  • Prospective Patients
* Sequential patients implanted with a CryoValve SG Pulmonary Human Heart Halve as a Ross or RVOT reconstruction after FDA 510(k) clearance in February 2008 at selected institutions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who have had a CryoValve SG Pulmonary Human Heart Valve implanted in the pulmonary position for right ventricular outflow tract (RVOT) reconstruction or as part of the Ross procedure at selected institutions.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Capps, MS, Study Director — CryoLife, Inc.
Locations (8):
- United States (8):
  - Arizona Pediatric Cardiology Consultants, Phoenix, Arizona
  - Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Oklahoma University Health and Sciences Center, Oklahoma City, Oklahoma
  - Cardiothoracic and Vascular Surgeons and Austin Heart, Austin, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Brown JW, Elkins RC, Clarke DR, Tweddell JS, Huddleston CB, Doty JR, Fehrenbacher JW, Takkenberg JJ. Performance of the CryoValve SG human decellularized pulmonary valve in 342 patients relative to the conventional CryoValve at a mean follow-up of four years. J Thorac Cardiovasc Surg. 2010 Feb;139(2):339-48. doi: 10.1016/j.jtcvs.2009.04.065. PMID 20106397
- [Background] Konuma T, Devaney EJ, Bove EL, Gelehrter S, Hirsch JC, Tavakkol Z, Ohye RG. Performance of CryoValve SG decellularized pulmonary allografts compared with standard cryopreserved allografts. Ann Thorac Surg. 2009 Sep;88(3):849-54; discussion 554-5. doi: 10.1016/j.athoracsur.2009.06.003. PMID 19699910
- [Background] Hawkins JA, Hillman ND, Lambert LM, Jones J, Di Russo GB, Profaizer T, Fuller TC, Minich LL, Williams RV, Shaddy RE. Immunogenicity of decellularized cryopreserved allografts in pediatric cardiac surgery: comparison with standard cryopreserved allografts. J Thorac Cardiovasc Surg. 2003 Jul;126(1):247-52; discussion 252-3. doi: 10.1016/s0022-5223(03)00116-8. PMID 12878962

RESULTS

PARTICIPANT FLOW:
Groups:
- Retrospective Patients: Retrospective Patients: These patients had the CryoValve SG Pulmonary Valve implanted prior to the February 2008 clearance of the valve.
Period: Overall Study
Arm/Group | Retrospective Patients | Prospective Patients
Started | 80 | 60
Completed | 80 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retrospective Patients | Prospective Patients | Total
Number analyzed (Participants) | 80 | 60 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 66 | 33 | 99
  Between 18 and 65 years | 14 | 26 | 40
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (14.1) | 26.2 (21.1) | 20.2 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 16 | 43
  Male | 53 | 44 | 97
Region of Enrollment [Number; unit: participants]
  United States | 80 | 60 | 140

OUTCOME MEASURES:

1. Primary Outcome: Hemodynamic Performance
Description: Peak Pulmonary Gradient Mean Pulmonary Gradient
Time Frame: Most Recent follow-up (average of 3-6 years post implant)
Population: The number of participants was limited to those participants with a hemodynamic measurement provided. Therefore, the total number in each group is less than the total participants in each group.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Retrospective Ross | Prospective Ross | Retrospective Right Ventricular Outflow Tract (RVOT) | Prospective RVOT
Number analyzed (Participants) | 25 | 39 | 47 | 19
mmHg
  Peak Pulmonary Gradient | 22.2 (16.0) | 13.5 (10.9) | 21.2 (11.4) | 21.9 (12.1)
  Mean Pulmonary Gradient | 12.1 (8.3) | 7.5 (5.7) | 12.3 (6.5) | 11.7 (6.7)

2. Primary Outcome: Hemodynamic Performance
Description: Pulmonary Insufficiency Grade
Time Frame: Most Recent Follow-up (average of 4 to 6 years post implant)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Retrospective Ross | Prospective Ross | Retrospective RVOT | Prospective RVOT
Number analyzed (Participants) | 27 | 39 | 48 | 19
participants
  None | 6 | 12 | 8 | 3
  Trivial | 6 | 18 | 14 | 13
  Mild | 10 | 6 | 12 | 2
  Moderate | 2 | 1 | 10 | 1
  Moderate-Severe | 1 | 1 | 1 | 0
  Severe | 0 | 1 | 3 | 0

3. Primary Outcome: Safety Assessment
Description: Evaluation of the following adverse events
  * Mortality (all cause and valve-related)
  * Reoperation/reintervention
  * Explant
  * Endocarditis
  * Structural valve deterioration (defined as >40 mmHg peak pulmonary gradient or >30 mmHg mean pulmonary gradient or moderately severe to severe pulmonary insufficiency)
  * Thrombosis
  * Thromboembolism (pulmonary embolism)
  * Non-structural dysfunction
  * Perivalvular leak
  * Bleeding
  * Hemolysis
  * Calcification
Time Frame: Since Implant of the Valve to a Maximum of 13.0 years
Measure: Number; unit: percentage of patients
Groups:
- Ross Patients: Retrospective and Prospective Patients that had the CryoValve SG Pulmonary Human Heart Valve implanted as a part of the Ross Procedure
- RVOT Reconstruction Patients: Retrospective and Prospective Patients that had the CryoValve SG Pulmonary Human Heart Valve implanted for RVOT reconstruction procedures
Arm/Group | Ross Patients | RVOT Reconstruction Patients
Number analyzed (Participants) | 68 | 72
percentage of patients
  10-Year Freedom from Mortality | 84 | 97
  10-Year Freedom from Valve-Related Mortality | 100 | 100
  10-Year Freedom from Reoperation/Reintervention | 100 | 81
  10-Year Freedom from Explant | 100 | 88
  10-Year Freedom from Endocarditis | 100 | 96
  10-Year Freedom from SVD | 74 | 52
  10-Year Freedom from Thrombosis | 100 | 100
  10-Year Freedom from Thromboembolism | 100 | 100
  10-Year Freedom from Non-structural Dysfunction | 100 | 100
  10-Year Freedom from Perivalvular Leak | 100 | 100
  10-Year Freedom from Bleeding | 96 | 96
  10-Year Freedom from Hemolysis | 100 | 100
  10-Year Freedom from Calcification | 80 | 63

ADVERSE EVENTS:
Time Frame: Since Implant of the Valve to a Maximum of 13 years
Description: Other Adverse Events were not collected
Arm/Group | Ross Patients | RVOT Reconstruction Patients
Serious Adverse Events (participants affected / at risk) | 5/68 | 11/72
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ross Patients (N=68) | RVOT Reconstruction Patients (N=72)
Mortality (Cardiac disorders) | 5 | 2
Explant (Cardiac disorders) | 0 | 4
Reoperation/Reintervention (Cardiac disorders) | 0 | 7
Endocarditis (Cardiac disorders) | 0 | 2
Bleeding (Cardiac disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can not publish any results or data arising from the study except with the institution's approval and sponsor's written consent.